CLINICAL TRIAL: NCT03601520
Title: Mechanisms of Pulmonary Diffusion Limitation in Systemic Sclerosis
Acronym: DL-SSc
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, MD, Pulmonary Function Lab Director, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: IRCCS-SSc-2018
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Diffusion Limitation of Pulmonary Gas Exchange in Systemic Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was designed to test the hypothesis that, irrespective of the degree of interstiaI lung disease and/or pulmonary arterial hypertension, the combined measurement of lung diffusing capacity for nitric oxide and carbon monoxide, might be useful to provide a mechanistic interpretation of changes of diffusion subcomponents in systemic sclerosis (SSc).

DETAILED DESCRIPTION:
In systemic sclerosis (SSc) the impairment of lung function is generally inferred from measurements of forced vital capacity (FVC) and standard lung diffusing capacity for carbon monoxide (DLCO). However, FVC measurement does not provide an accurate estimate of lung restriction and DLCO does not allow separate the alveolar membrane (DMCO) from erythrocyte (DeCO) diffusive conductance for CO. Previous studies have shown that DMCO and DeCO may change irrespective of overt intersitial lung disease (ILD) and/or pulmonary arterial hypertension (PAH). These changes may be consistent with a limitation of alveolar-capillary erythrocyte recruitment which impairs DM.This study was designed to test the hypothesis that, irrespective of the degree of ILD and/or PAH, combined DLNO-DLCO measurement might be useful to provide a mechanistic interpretation of DM and De changes in SSc.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilling the 2013 American College of Rheumatology/European League Against Rheumatism criteria for a definite diagnosis of SSc with a total score ≥9

Exclusion Criteria:

* unstable subjects and/or who have suffered from respiratory exacerbations in the previous 4-wk

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SSc patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Lung diffusing capacity for nitric oxide | 2 hours
  Alveolar-capillary gas exchange

REFERENCES:
- [Background] Barisione G, Bacigalupo A, Brusasco C, Scanarotti C, Penco S, Bassi AM, Lamparelli T, Garlaschi A, Pellegrino R, Brusasco V. Mechanisms for reduced pulmonary diffusing capacity in haematopoietic stem-cell transplantation recipients. Respir Physiol Neurobiol. 2014 Apr 1;194:54-61. doi: 10.1016/j.resp.2014.01.018. Epub 2014 Feb 1. PMID 24495442
- [Background] Barisione G, Brusasco C, Garlaschi A, Baroffio M, Brusasco V. Lung diffusing capacity for nitric oxide as a marker of fibrotic changes in idiopathic interstitial pneumonias. J Appl Physiol (1985). 2016 May 1;120(9):1029-38. doi: 10.1152/japplphysiol.00964.2015. Epub 2016 Feb 18. PMID 26893034
- [Derived] Barisione G, Garlaschi A, Occhipinti M, Baroffio M, Pistolesi M, Brusasco V. Value of lung diffusing capacity for nitric oxide in systemic sclerosis. Physiol Rep. 2019 Aug;7(13):e14149. doi: 10.14814/phy2.14149. PMID 31264386